> Protocol No: RD.03.SPR.112075 Statistical Analysis Plan Page 1 of 37

# EXPLORATORY STUDY TO EVALUATE THE SAFETY AND EFFICACY OF CD10367 IN SUBJECTS WITH PSORIASIS

STATISTICAL ANALYSIS PLAN RD.03.SPR.112075 Project 315 EudraCT Number 2016-002774-12

Version of 09/03/2017

| Author: | PPD | |
|-----------|-------------------------------------------|------|
| | PPD Galderma R&D – Biostatistician | Date |
| | PPD | |
| Reviewer: | | |
| | PPD | |
| | Galderma R&D – Expert Statistician Senior | |

# LIST OF ABBREVIATIONS AND DEFINITIONS OF TERMS

| Abbreviations | Terms |
|---------------|----------------------------------------------|
| AEs | Adverse events |
| ATC | Anatomical Therapeutic Chemical |
| AUC | Area Under Curve |
| BLQ | Below Limit of Quantification |
| CV | Coefficient of variation |
| EGFR | Epidermal Growth Factor Receptor |
| ERK | Extracellular signal – Regulated Kinases |
| ET | Early Termination |
| FU | Follow Up |
| IHC | Immuno Histo Chemistry |
| ITT | Intent-To-Treat |
| Ln | Logarithmic |
| LOCF | Last Observation Carried Forward |
| LOQ | Limit Of Quantification |
| MedDRA | Medical Dictionary for Regulatory Activities |
| N | Number |
| NA | Not Applicable |
| CCI | |
| PK | PharmacoKinetic |
| PP | Per protocol |
| PT | Preferred Term |
| R&D | Research & Development |
| SAEs | Serious Adverse Events |
| SAS | Statistical Analyses System |
| SD | Standard deviation |
| SOC | System Organ Class |
| TSS | Total Sum Score |
| WHO | World Health Organization |

# **TABLE OF CONTENTS**

| 1. | STUDY OBJECTIVES6 |
|---|---|
| 2. | STUDY DESIGN6 |
| 3. | EFFICACY AND SAFETY ASSESSMENT8 |
| 4. | EFFICACY AND SAFETY VARIABLES9 |
| 4.1. | Efficacy variables9 |
| 4.2. | Safety variables |
| CCI | |
| 5. | POPULATIONS ANALYZED |
| 5.1. | The Intent-to-treat (ITT) population11 |
| <b>5.2.</b> | The Per-Protocol (PP) efficacy population12 |
| 5.3. | The Safety population12 |
| 7. | STATISTICAL METHODS AND DATA CONSIDERATIONS |
| 7.1. | Study subjects14 |
| 7.1.1 | Disposition of subjects14 |
| 7.1.2 | Protocol deviations |
| 7.2. | Efficacy analysis14 |
| 7.2.1. | Data sets analyzed14 |
| 7.2.2. | Demographic characteristics |
| 7.2.3 | Medical history, previous and concomitant therapies, medical and surgical procedures |
| 7.2.4. | Compliance |
| 7.2.5. | Efficacy analysis |
| 7.2.5. | Primary and secondary efficacy analysis |

| Statisti<br>Page 4 | cal Analysis Plan<br>of 38 |
|--------------------|-----------------------------------------------------|
| 7.2.6. | Statistical and analytical issues16 |
| 7.2.6.1 | Adjustment for covariates |
| 7.2.6.2 | Handling of dropouts or missing data |
| 7.2.6.3 | Interim analyses and data monitoring |
| 7.2.6.4 | Multicenter studies |
| 7.2.6.5 | Multiple comparison/multiplicity |
| 7.2.6.6 | Use of an efficacy subset of patients |
| 7.2.6.7 | Active-Control studies intended to show equivalence |
| 7.2.6.8 | Examination of Subgroups |
| 7.3. | Safety analysis |
| 7.3.1. | Extent of exposure17 |
| 7.3.2. | Local tolerance17 |
| 7.3.3. | Adverse events17 |
| 7.3.4. | Physical examination, vital signs17 |
| 7.3.5. | Ophthalmic examination17 |
| 7.3.6. | 12-lead electrocardiogram18 |
| CCI | |
| 7.3.8. | Laboratory parameters18 |
| CCI | |
| 7.4.1. | Plasma concentration |
| CCI | |
| 7.5. | Analysis visit definition |
| 8. | CHANGES FROM THE PROTOCOL ANALYSIS PLAN |
| 9. | TABLES, FIGURES AND GRAPHS20 |
| 9.1. | Study subjects20 |
| 9.2. | Efficacy analyses |
| 9.2.1. | Subjects characteristics20 |
| 9.2.2. | Baseline characteristics21 |
| 9.2.3. | Primary and secondary efficacy criteria22 |
| 9.3. | Safety analyses |
| 9.3.1. | Extent of exposure |
| 9.3.2. | Local tolerance |
| 9.3.3. | Adverse events31 |
| 9.3.4. | Vital Signs, Physical Findings32 |

| Protoco | l No: RD.03.SPR.112075 | |
|-----------|------------------------|----|
| Statistic | cal Analysis Plan | |
| Page 5 | of 38 | |
| 9.3.5. | Laboratory Parameters | 34 |
| 9.4. | Graphs | 35 |
| CCI | | |

#### 1. STUDY OBJECTIVES

The primary objective is to evaluate, in a modified Dumas-Scoltz psoriasis mini-zone test, the safety and efficacy of CD10367 solution at 1% and 3% after a three weeks treatment period of once daily application.



#### 2. STUDY DESIGN

Phase IIa.

This is an exploratory, single-centre (France), investigator blinded, randomized, controlled, intraindividual study (Dumas-scholtz design).

Approximately 40 male or female of at least 18 and up to 70 years old suffering from stable plaque psoriasis vulgaris will be screened to randomize 24 subjects.

The subjects will be screened within 3 weeks prior to the pre-treatment period of up to 2 weeks, followed by a treatment period of 3 weeks and a follow-up period of 1 week.

During the pre-treatment period, the subject will apply a keratolytic product at home twice a day on the selected plaques defined by the investigator.

(tube 50ml) with 50% of urea and 2% of salicylic acid (other components: serine, histidine, glycenin, protease, fragrance free and paraben free) will be used as the keratolytic agent. On these target areas, the desquamation will be controlled by the dermatologist and if the scaling's score is 0 or 1 (none or mild), the subject will be enrolled.



Statistical Analysis Plan


A final visit at Day 19 (or early termination visit if any) will be performed to evaluate safety and efficacy of the treatments,

CC

The study is expected to last approximately 5 months from the first subject included in the study to the last visit of the last subject. The total maximum study duration for one subject will be 9 weeks.


# 3. EFFICACY AND SAFETY ASSESSMENT

| | Screening period | | | | | | Tre | Follow-up period | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Up to 3 weeks before | | | Week 1 | Week 2 | | | | Week 3 | | | Week 4 to 5 | | |
| | pre-treatment period | treatment period | D1 | D2 &D3 | D4 | D5 | D8 | D9 & D10 | D11 | D12 | D15 | D16&D17&D18 | Final visit D19 /ET | D26 +/- 2 |
| Informed Consent Form | X | | | | | | | | | | | | | |
| Demographics and Medical history | Х | | | | | | | | | | | | | |
| Previous treatments and procedures | Х | | | | | | | | | | | | | |
| Physical examination | Х | | | | | | | | | | | | Х | |
| Vital signs | Х | | Х | | | | | | | | | | Х | |
| ECG | > | ( b | | | | | | | | | | | Х | |
| Ophthalmic examination | > | <b>(</b> b | | | | | | | | | | | Х | |
| Inclusion Criteria and Exclusion Criteria | Х | | Х | | | | | | | | | | | |
| Selection of target sites | Х | | Х | | | | | | | | | | | |
| Urinalysis | Х | | | | | | | | | | | | Х | |
| Safety tests Blood sampling | X | | | | | | | | | | | | Х | |
| Randomization | | | Х | | | | | | | | | | | |
| Local Tolerance ° | | | | D2 only | Χ | | Χ | | Х | | Х | | Х | |
| Individual clinical scores | Х | | Х | | Χ | | Χ | | Х | | Х | | Х | |
| Clearing score | | | | | Χ | | Χ | | Х | | Х | | Х | |
| Keratolytic product application of selected plaque at home daily | | X | | | | | | | | | | | | |
| Products application | | | Χ | Х | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | | |
| CCI | 1 | ı | | • | ı | 1 | 1 | | 1 | | 1 | | I | |
| PK blood sampling | | | | | | Χ | | | | | | | X | X |
| CCI | | | | | | | | | | | | | | |
| Concomitant treatments and Procedures | Х | Х | Χ | Х | Χ | Χ | Χ | Х | Χ | Χ | Χ | Х | Х | Х |
| Adverse events d | Х | Х | Х | Х | Χ | Χ | Χ | Х | Х | Х | Χ | Χ | Х | Х |
| Exit form e | | | | | | | | | | | | | Χf | Х |

a. if the scaling score did not reach 0 or 1 after 1 week of pre-treatment, the pre-treatment period can be extended to 2 weeks, otherwise the subjects will start D1 visit immediately. b ECG and ophthalmic exams should be done as close as possible to baseline visit. c Local tolerance of the concerned zone must be taken at any visit in case of AE in a treatment zone. d Adverse Events have to be collected from the ICF signature. e Exit form should be signed after subject data collection has been completed. f Exit form should be completed at ET visit only if no follow-up visit is planned (discontinuation)

Statistical Analysis Plan


#### 4. EFFICACY AND SAFETY VARIABLES

# 4.1. Efficacy variables

Primary clinically efficacy criteria

Area Under the Curve (AUC) from Day 1 to Day 19 of Total Sum Score (TSS) (sum of erythema, scaling and induration scores).

Secondary clinically efficacy criteria

- AUC of individual clinical scores (erythema, scaling and induration) from Day 1 to Day 19.

Erythema is scored on the following 5-point scale:

| 0 | None | No detectable erythema. |
|---|-------------|--------------------------------------|
| 1 | Mild | Slight pinkness present |
| 2 | Moderate | Definite redness, easily recognized. |
| 3 | Severe | Intense redness |
| 4 | Very Severe | Very intense redness |

<u>Scaling</u> is scored on the following 5-point scale:

| 0 | None | No shedding |
|---|---|---|
| 1 | Mild | Barely perceptible shedding, noticeable only on light scratching or rubbing. |
| 2 | Moderate | Obvious but not profuse shedding |
| 3 | Severe | Heavy scale production |
| 4 | Very Severe | Very thick scales |

<u>Induration</u> is scored on the following 5-point scale:

| 0 | None | Normal skin thickness. No elevation of skin |
|---|---|---|
| 1 | Mild | Barely perceptible elevation (by touching) of the psoriasis plaques. |
| 2 | Moderate | Obvious elevation above the normal skin level; moderate thickening |
| 3 | Severe | Definite thick elevation above normal skin level |
| 4 | Very Severe | Very thick elevation |

- TSS at each visit (screening, end of pre-treatment period for Z1 and Z2, day 1, day 4, day 8, day 11, day 15 and day 19) and TSS percent change from baseline;
- Erythema, scaling and induration score at each visit: screening, end of pretreatment period for Z1 and Z2, day 1, day 4, day 8, day 11, day 15 and day 19) and their change from day 1;
- Success rate (defined as a clearing score of 0 or 1) at each evaluation visit (day 4, day 8, day 11, day 15 and day 19) and the time to first success.

Statistical Analysis Plan


The clearing score is defined as:

| 0 | Complete clearing | No scaling and no infiltration even on palpation. Post inflammatory hypo- or hyperpigmentation may be present. |
|---|---|---|
| 1 | Almost clear | Residual erythema with some induration/ infiltration (not clinically visible but palpable) without scaling, or residual erythema and residual scaling with no infiltration. |
| 2 | Unchanged | Unchanged or less than almost clear. |

The time to partial clearing (clearing score of 0 or 1) is defined as:

| 0 | No Success at any day |
|---|----------------------------------|
| 1 | Success at Day 19 and not before |
| 2 | Success at Day 15 and not before |
| 3 | Success at Day 11 and not before |
| 4 | Success at Day 8 and not before |
| 5 | Success at Day 4 and not before |

Only the earliest day of success will be considered in defining the time to partial clearing, independently of the subsequent days.



# 4.2. Safety variables

- Local tolerance (irritation, stinging/burning, pruritus) twice weekly using a 4-point scale for each mini-zone:

| Irritation | Skin irritati | Skin irritation Assessment |
|---|---|---|
| 0 | None: | No signs of irritation |
| 1 | Mild: | Slight signs of irritation |
| 2 | Moderate: | oderate signs of irritation: Obvious increase in redness as compared to the n-treated surrounding area |
| 3 | Severe: | Severe signs of irritation |
| Stinging/ Burning | Prickling pa | nin sensation |
| 0 | None: | No stinging/burning |
| 1 | Mild: | Slight warm, tingling/stinging sensation; not really bothersome |
| 2 | Moderate: | Definite warm, tingling/stinging sensation that is somewhat bothersome |
| 3 | Severe: | Hot, tingling/stinging sensation that causes severe discomfort |
| Pruritus | Itch sensati | on |
| 0 | None: | No itching |
| 1 | Mild: | Itching is noticeable but not really bothersome |

Statistical Analysis Plan


| 2 | Moderate: | Definite itching that is somewhat bothersome |
|---|---|---|
| 3 | Severe: | Marked itching, urge to scratch and causes definite discomfort |

- Incidence and multiplicity of Adverse Events (from informed consent signature to the end of the study);
- Ophtalmic examination at screening and day 19/ET
- Physical examination at screening and day 19/ET;
- Vital signs performed after 5 minutes rest in the sitting position (systolic blood pressure, diastolic blood pressure, pulse rate, vital signs evaluation) at screening, baseline and day 19/ET;
- 12-lead electrocardiogram during the screening period and at day 19/ET;
- Blood samplings for laboratory safety tests (haematology and blood chemistry) at screening and day 19/ET (Virology will be performed only at screening);
- Urinalysis at screening and day 19/ET;



# 5. POPULATIONS ANALYZED

# 5.1. The Intent-to-treat (ITT) population

The ITT Population is defined as comprising all subjects who are randomized.


# 5.2. The Per-Protocol (PP) efficacy population

This population will consist of ITT subjects, except some subjects considered as not evaluable due to major deviations from protocol.

Major deviations will be defined after data entry and before breaking the treatment blind, and may include: inclusion criteria not respected, interfering therapy, protocol deviation, poor compliance to study treatment administration or protocol requirements, unblinding. The decision on determining whether a subject is excluded from the per-protocol (PP) population will be made during the blind review meeting.

If no patient has a major deviation, PP efficacy population will be the same as ITT population, and results will be presented on the ITT population only.

# 5.3. The Safety population

Safety population corresponds to all subjects who received at least once the study treatment during the treatment period.

In case of identical populations, only one safety population will be used for the analysis.





# 7. STATISTICAL METHODS AND DATA CONSIDERATIONS

SAS® version 9.3 will be used for the analysis. Graphics will be performed on SAS.

The categorical variables will be summarized by frequency and percentage for each response category (N, %). The continuous variables will be summarized using means, medians, minimum, maximum, and standard deviations.


# 7.1. Study subjects

# 7.1.1. Disposition of subjects

Subject disposition will be summarized in the ITT population.

Normal completion as well as early discontinuation will be summarized using frequency distribution (n, %). All early discontinuations will be detailed in a subject-by-subject listing.

#### 7.1.2. Protocol deviations

All protocol deviations, including the decisions regarding major/minor protocol deviations, will be documented in the blind data review meeting and entered into a dataset.

Subjects with major protocol deviations will be excluded from the PP population.

Major protocol deviations will be summarized using frequency distribution (n, %) and will be detailed in a subject-by-subject listing.

# 7.2. Efficacy analysis

# 7.2.1. Data sets analyzed

Number of subjects included in each population (ITT population, PP population, safety population, CCI) will be summarized.

# 7.2.2. Demographic characteristics

Frequency distribution (n, %), for qualitative criteria, will be used.

Usual descriptive statistics (n, mean, standard deviation, median, min, max), for quantitative criteria, will be used.

Analysis will be performed on ITT population and PP population (if the number of patients is too different).

# 7.2.3. Medical history, previous and concomitant therapies, medical and surgical procedures

Medical history will be defined as any disease present before the Screening visit.

Frequency distribution of subjects with previous or/and concomitant disease(s) will be tabulated. Previous and concomitant therapies will be coded using the World Health Organization (WHO) Drug Dictionary (version v032015).

Previous therapies are defined as therapies stopped within the 6 months preceding the screening visit. Frequency distribution of subjects with at least one previous therapy will be tabulated by Anatomical Therapeutic Chemical (ATC) classification.

Concomitant therapies are defined as any ongoing therapies at the time of the screening visit, and any new therapies started or changed since the screening visit.

Frequency distribution of subjects with at least one concomitant therapy will be tabulated by ATC classification.

Previous and concomitant procedures will be coded using the Medical Dictionary for Regulatory Activities (MedDRA version 18.0).

Previous procedures are defined as procedures stopped within 6 months preceding the screening visit.

Statistical Analysis Plan


Frequency distribution of subjects with at least one previous procedure will be tabulated (n, %) by preferred term.

Concomitant procedures are defined as any ongoing procedures at the time of the screening visit, and any new procedures started or changed since the screening visit.

Frequency distribution of subjects with at least one concomitant procedure will be tabulated (n, %) by preferred term.

### 7.2.4. Compliance

extreme cream will be applied at home by the subject twice daily, up to 2 weeks before the treatment period upon the judgment of the dermatologist. The scaling score should be 0 or 1 when the subject is enrolled.

All applications during the treatment period will be performed by a person from the investigational team at the study centre, once daily during 3 weeks, 5 days a week except for the third week, for a total of 14 applications.

Subjects with a low compliance will be excluded from PP population during the data review.

# 7.2.5. Efficacy analysis

# 7.2.5.1 Primary and secondary efficacy analysis

Descriptive statistics will be done on observed cases for PP and ITT populations.

The Area Under the Curve (AUC) will be calculated from Day 1 (before application) to Day 19 by subject and by treatment/pre-treatment on the Z1-Z6 mini-zone, using the trapezoidal rule on ITT and PP population.

Dates of theorical visit will be used to perform AUC.

AUC of TSS will be submitted to an analysis of variance including subject and treatment/pre-treatment as factors in the model,

AUC of individual clinical scores (erythema, scaling and induration) will be submitted to the same variance analysis.

TSS and TSS percent change from day 1 will be descriptively summarized by visit, as the individual score of erythema, scaling and induration and their respective change from day 1. The analysis will be performed on PP population and ITT population (baseline and Endpoint/LOCF) Success will be presented in frequency tables (N,%) by treatment/pre-treatment and by visit.

The time to first success will be summarized by treatment/pre-treatment.




# 7.2.6. Statistical and analytical issues

# 7.2.6.1 Adjustment for covariates

Adjustments to baseline value, i.e., day 1 will be considered in the calculation of change and percent change.

# 7.2.6.2 Handling of dropouts or missing data

For evaluation by visit, on ITT population, a last visit named "Endpoint/LOCF" containing the last observation carried forward (LOCF) will be created.

For Area Under the Curves (of the TSS or for each individual clinical score), no imputation for missing assessment will be done and calculations will be done on observed data, nevertheless for the subjects who terminated earlier, the Final Visit will be imputed to the closest theoretical visit of the protocol.

For patients who have individual score assessments on unscheduled day, closest theoretical visit of the protocol will be used, for each evaluation overtime and AUC.

# 7.2.6.3 Interim analyses and data monitoring

Not Applicable (NA)

7.2.6.4 Multicenter studies

NA

# 7.2.6.5 Multiple comparison/multiplicity

| CCI | |
|---------------|-----------------------------------------------------|
| 7.2.6.6<br>NA | Use of an efficacy subset of patients |
| 7.2.6.7<br>NA | Active-Control studies intended to show equivalence |
| 7.2.6.8<br>NA | Examination of Subgroups |


# 7.3. Safety analysis

All safety data will be summarized based on the safety population.

# 7.3.1. Extent of exposure

Number of days of keratolytic during the pre-treatment period in zone 1 and 2 will be summarized.

Study product application will be presented by treatment/pre-treatment and by visit.

Number of study products applications will be summarized by treatment/pre-treatment.

# 7.3.2. Local tolerance

Local individual signs/symptoms (irritation, skinging/burning, pruritus) in term of frequency distribution and in quantitative description and the worst score (from Day 2 to Day 19/ET) over time of each individual sign/symptom will be calculated by study product.

#### 7.3.3. Adverse events

Adverse Events will be tabulated by study treatment/pre-treatment and in overall.

Occurrence of adverse events will be separated in two periods: the pre-treatment period from the beginning of the pre-treatment period to day 1 excluded, and the treatment period from the date of first application of study drugs to the end of the study.

For the pre-treatment period, only a table with the overview of the adverse events and a listing of the adverse events during this period will be performed.

For the treatment period, Adverse Events (AE) will be tabulated in frequency tables by System Organ Class (SOC) and Preferred Term (PT) based on MedDRA version 18.0. Additional summary tables will be provided for Adverse Events that are considered serious (SAEs), related to study product, related to protocol procedure, related to the study (study product and/or protocol procedure), Adverse Events of special interest, and Adverse Events leading to discontinuation.

Due to the intra-individual study design and whenever possible (known from CRF) AE will be imputed to the treated area, when not possible then the AE will be imputed to all treated zones.

AEs with an onset prior to the pre-treatment period will be listed separately.

# 7.3.4. Physical examination, vital signs

Physical examination and vital signs evaluation will be summarized by visit using frequency tables (Normal/Abnormal and not clinically significant/Abnormal and clinically significant). Shift table will be tabulated.

Systolic blood pressure, diastolic blood pressure and pulse rate will be summarized by visit in quantitative manner. Change from baseline will be calculated.

# 7.3.5. Ophthalmic examination

Ophthalmic examination will be summarized by visit using frequency tables (Normal/Abnormal and not clinically significant/Abnormal and clinically significant).


Shift table will be tabulated.

# 7.3.6. 12-lead electrocardiogram

Results of 12-lead electrocardiogram will be summarized by visit using frequency tables (Normal/Abnormal and not clinically significant/Abnormal and clinically significant). Shift table will be tabulated.

QTc interval and change from screening will be also summarized by visit.



# 7.3.8. Laboratory parameters

Each hematology and biochemistry parameter will be subject to quantitative and qualitative analyses at screening and at day 19/ET.

Quantitative values in standard units will be summarized at screening and at Day 19/ET, as well as change from screening.

Frequency of subjects with low, normal, high values with respect to normal range will be summarized at screening and at day 19/ET.

Shift tables will be displayed presenting data at screening and at day 19/ET.

Each urinalysis parameter will be subject to qualitative analyses at screening and at day 19/ET. Shift tables will also be displayed.

In case of urinalysis parameter in quantitative manner, results will be presented by summary statistics.



#### 7.4.1. Plasma concentration

Raw values of concentration of CD10367 will be summarized with geometric mean, arithmetic mean, standard deviation (SD), coefficient of variation (CV), median, minimum and maximum values by visit (day 5; day 19/ET and day 26).

Logarithmic values (ln) of concentration of CD10367 will be summarized with mean, standard deviation, median, minimum and maximum value by visit.





#### 7.5. **Analysis visit definition**

NA

#### 8. CHANGES FROM THE PROTOCOL ANALYSIS PLAN

NA


# 9. TABLES, FIGURES AND GRAPHS

# 9.1. Study subjects

Table. Enrollment by Center

Table. Subjects who discontinued treatment and reason for discontinuation

Table. Major protocol deviations

# 9.2. Efficacy analyses

# 9.2.1. Subjects characteristics

Table. Data sets analyzed

# Table. Demographic data - ITT population

Including age (as quantitative data and by class 18-64, 65-84 and >=85), gender, race, phototype, subject of childbearing potential.

#### Table. Medical history – ITT population

Including duration of psoriasis and relevant or major illnesses present before the screening visit.

Table. Previous therapies by ATC term-ITT population

Table. Previous procedures by preferred term – ITT population

Table. Concomitant therapies by ATC term - ITT population

Table. Concomitant procedures by preferred term – ITT population


# 9.2.2. Baseline characteristics

# Table. Target location – ITT population

| | CD10367 placebo<br>pre-treated | CD10367 3%<br>pre-treated | CD10367<br>placebo | CD10367 1% | CD10367 3% | Betneval 0.1% | Overall |
|---|---|---|---|---|---|---|---|
| N<br>Elbows<br>Knees | n(%)<br>n(%) | | | | | | |

# Table. Target location - PP population

# Table. Pre-treatment clinical scores in mini-zones Z1 and Z2 – ITT population

| | | CD10367 placebo<br>pre-treated | CD10367 3%<br>pre-treated | Overall |
|---|---|---|---|---|
| Erythema | N | <del>-</del> | | |
| | 2 | | | |
| | 3 | | | |
| | 4 | | | |
| | Mean | | | |
| | SD | | | |
| | Median | | | |
| | (Min,Max) | | | |
| Scaling | N | | | |
| | 0 | | | |
| | 1 | | | |
| | Mean | | | |
| | SD | | | |
| | Median | | | |
| | (Min,Max) | | | |
| Induration | | | | |
| TSS | | | | |

Table. Pre-treatment clinical scores in mini-zones Z1 and Z2 - PP population

Table. Baseline clinical scores in mini-zones Z1 to Z6 – ITT population


Baseline corresponds to week 1 day 1.

# Table. Baseline clinical scores in mini-zones Z1 to Z6 – PP population

Baseline corresponds to week 1 day 1.

# 9.2.3. Primary and secondary efficacy criteria

# Table. AUC of TSS - Treatment period - PP and ITT population

| | | CD10367 | CD10367 | CD10367 placebo | CD10367 1% | CD10367 3% | Betneval 0.1% |
|---|---|---|---|---|---|---|---|
| | | placebo | 3% | | | | |
| | | pre-treated | pre-treated | | | | |
| AUC of TSS (PP) | N | | | | | | |
| | Mean | | | | | | |
| | SD | | | | | | |
| | Median | | | | | | |
| | (Min,Max) | | | | | | |
| AUC of TSS (ITT) | N | | | | | | |
| | Mean | | | | | | |
| | SD | | | | | | |
| | Median | | | | | | |
| | (Min,Max) | | | | | | |

# Table. Analysis of variance for AUC of TSS – Treatment period - PP population

| | | LSmean(SE) | p-value* |
|---------------|--------------------------------|------------|----------|
| Model Effects | Patient | - | |
| Treatment | CD10367 placebo pre-treated | | |
| Treatment | CD10367 3% pre-treated | | |
| Contrast | <br>CD10367 placebo – Betneval | | |
| | ••• | | |
| CCI | | | |


Table. AUC of erythema - Treatment period - PP and ITT population

Table. Analysis of variance for AUC of erythema – Treatment period - PP population

Table. AUC of scaling – Treatment period - PP and ITT population

Table. Analysis of variance for AUC of scaling – Treatment period - PP population

Table. AUC of induration – Treatment period - PP and ITT population

Table. Analysis of variance for AUC of induration – Treatment period - PP population

Table. TSS and TSS percent change from day 1 – PP population

| TSS | | CD10367 | CD10367 3% | CD10367 | CD10367 1% | CD10367 | Betneval |
|---|---|---|---|---|---|---|---|
| | | placebo | pre-treated | placebo | | 3% | 0.1% |
| | | pre-treated | | | | | |
| Screening | N | | | | | | |
| | Mean | | | | | | |
| | SD | | | | | | |
| | Median | | | | | | |
| | (Min,Max) | | | | | | |
| End of pre-treatment period* | | | | | | | |
| Day 1, Day 4 | N | | | | | | |
| | Mean | | | | | | |
| | SD | | | | | | |
| | Median | | | | | | |
| | (Min,Max) | | | | | | |
| Percent change from Day 1 at Day 4 | N | | | | | | |
| | Mean | | | | | | |
| | SD | | | | | | |
| | Median | | | | | | |
| | (Min,Max) | | | | | | |
| Day 8, Day 11, Day 15, Day 19 | N | | | | | | |
| Percent change from Day 1 at Day | <br>N | | | | | | |
| 8, Day 11, Day 15, Day 19 | 14 | | | | | | |
| inarformed only in 71 and 72 | ••• | | | | | | |

<sup>\*</sup>performed only in Z1 and Z2


Table. TSS and TSS percent change from day 1 – ITT population

ITT population and with only 2 visits: Day 1 and Endpoint/LOCF

Table. Erythema and change from day 1 – PP population

Table. Erythema and change from day 1 – ITT population

Table. Scaling and change from day 1 -PP population

Table. Scaling and change from day 1 –ITT population

Table. Induration and change from day 1 – PP population

Table. Induration and change from day 1 – ITT population

Table. Clearing score by visit – Treatment period - PP population

| Clearing score | | CD10367 placebo<br>pre-treated | CD10367 3%<br>pre-treated | CD10367 placebo | ••• | ••• |
|---|---|---|---|---|---|---|
| Day 4 | N | | | | | |
| | 0 | | | | | |
| | 1 | | | | | |
| | 2 | | | | | |
| | Mean | | | | | |
| | SD | | | | | |
| | Median | | | | | |
| | (Min,Max) | | | | | |
| Day 8, Day 11, Day 15, Day 19 | | | | | | |

# Table. Clearing score by visit – Treatment period - ITT population

Same table as above but on ITT population and with the additional visit Endpoint/LOCF


# Table. Success by visit – Treatment period - PP population

| Success | | CD10367<br>placebo<br>pre-treated | CD10367 3%<br>pre-treated | CD10367 placebo | <br> |
|---|---|---|---|---|---|
| Day 4 | N<br>No<br>Yes | | | | |
| Day 8, Day 11, Day 15, Day 19 | N<br>No<br>Yes | | | | |

# Table. Success by visit – Treatment period - ITT population

# Table. Time to first success - Treatment period - PP and ITT population

| Time to first success | | CD10367<br>placebo<br>pre-treated | CD10367 3%<br>pre-treated | CD10367 placebo | <br> |
|---|---|---|---|---|---|
| PP | N No success at any day Success at Day 19 and not before Success at Day 15 and not before Success at Day 11 and not before Success at Day 8 and not before Success at Day 4 and not before Mean SD Median (Min,Max) | • | | | |
| ITT | ••• | | | | |

Internally Approved 01-Feb-2019 Protocol No: RD.03.SPR.112075


Statistical Analysis Plan 



Internally Approved 01-Feb-2019 Protocol No: RD.03.SPR.112075


Statistical Analysis Plan 




# 9.3. Safety analyses

# 9.3.1. Extent of exposure

# Table. Pre-treatment duration of keratolytic product – Safety population

| | | CD10367 placebo | CD10367 3% |
|---|---|---|---|
| | | pre-treated | pre-treated |
| Number of days of keratolytic product applications | N | | |
| | 4 | | |
| | 5 | | |
| | 6 | | |
| | 7 | | |
| | N | | |
| | Mean | | |
| | SD | | |
| | Median | | |
| | (Min,Max) | | |


# Table. Study drug applications during the treatment period on mini-zones Z1 to Z6 - Safety population

| | | CD10367<br>placebo<br>pre-treated | CD10367 3%<br>pre-treated | CD10367 placebo | <br> |
|---|---|---|---|---|---|
| Day 1 | N | | | | |
| | No | | | | |
| | Yes | | | | |
| Day 2, 3 4, 5, 8, 9, 10, 11, 12, 15, 16, 17,18 | N | | | | |
| | No | | | | |
| | Yes | | | | |
| Day 2: reason for not applied | N Temporarily discontinued due to irritation Permanent discontinuation due to irritation Other | | | | |

# $Table.\ Number\ of\ applications\ during\ the\ treatment\ period\ on\ mini-zones\ Z1\ to\ Z6-Safety\ population$

| | CD10367 placebo | CD10367 3% | CD10367 placebo | ••• |
|-----------|-----------------|-------------|-----------------|-----|
| | pre-treated | pre-treated | | |
| N | | | | |
| 11 | | | | |
| 12 | | | | |
| 13 | | | | |
| Mean | | | | |
| SD | | | | |
| Median | | | | |
| (Min,Max) | | | | |


# 9.3.2. Local tolerance

#### Table. Irritation in term of continuous data

| Irritation | CD10367 placebo<br>pre-treated | CD10367 3%<br>pre-treated | CD10367 placebo | ••• | ••• | ••• |
|---|---|---|---|---|---|---|
| Day 2 | | | | | | |
| N | XX | XX | XX | XX | XX | XX |
| Mean±sd<br>Median<br>(Min,Max)<br>Day 3 | xx.x±xx.x<br>xx.x<br>(xx.x, xx.x) | xx.x±xx.x<br>xx.x<br>(xx.x, xx.x) | xx.x±xx.x<br>xx.x<br>(xx.x, xx.x) | xx.x±xx.x<br>xx.x<br>(xx.x, xx.x) | xx.x±xx.x<br>xx.x<br>(xx.x, xx.x) | xx.x±xx.x<br>xx.x<br>(xx.x, xx.x) |
| Day 19 | | | | | | |
| Day 19/ET | | | | | | |
| Follow-up | | | | | | |

0= None - 1=Mild - 2=Moderate - 3=Severe

# Table. Irritation in term of frequency distribution

| Irritation | | CD10367 placebo<br>pre-treated | CD10367 3%<br>pre-treated | CD10367 placebo | ••• |
|---|---|---|---|---|---|
| Day 2 | N<br>0- None | | | | |
| | 1- Mild | | | | |
| | 2- Moderate | | | | |
| | 3 – Severe | | | | |
| Day 2 | | | | | |

Table. Stinging /Burning in term of continuous data

Table. Stinging /Burning in term of frequency distribution

Table. Pruritus in term of continuous data

Table. Pruritus in term of frequency distribution

Table. Worst Score in term of frequency distribution

#### 9.3.3. Adverse events

- Table. Overview of adverse events during the pre-treatment period Safety population
- Table. Listing of adverse events during the pre-treatment period Safety population
- Table. Listing of adverse events prior the pre-treatment period Safety population

†Or listing if few AE.

- Table. Overview of adverse events during the treatment period Safety population
- Table †. Summary of adverse events by Preferred Term Safety population
- Table †. Summary of adverse events Related to the study drug by Preferred Term Safety population
- Table †. Summary of adverse events Related to the protocol procedure by Preferred Term Safety population
- Table †. Summary of adverse events Related to the study by Preferred Term Safety population
- Table . Summary of adverse events by System Organ Class and Preferred term Safety population
- Table †. Summary of adverse events Related to the study drug by System Organ Class and Preferred term Safety population
- Table †. Summary of adverse events Related to the protocol procedure by System Organ Class and Preferred term Safety population
- Table †. Summary of adverse events Related to the study by System Organ Class and Preferred term Safety population
- Table †. Summary of adverse events by severity by System Organ Class and by Preferred term Safety population
- Table †. Summary of adverse events Related to the study drug by severity by System Organ Class and by Preferred term Safety population
- Table †. Summary of adverse events Related to the protocol procedure by severity by System Organ Class and by Preferred term Safety population
- Table †. Summary of adverse events Related to the study by severity by System Organ Class and by Preferred term Safety population
- Table †. Summary of serious adverse events by System Organ Class and by Preferred term Safety population
- Table †. Summary of adverse events leading to discontinuation by System Organ Class and by Preferred term Safety population
- Table †. Summary of AESIs by System Organ Class and by Preferred term Safety population


# 9.3.4. Vital Signs, Physical Findings

# Table. Physical examination – Safety population

| | | Screening | DAY 19/ET |
|---|---|---|---|
| Physical examination | N | | |
| | Normal | | |
| | Abnormal and Not clinically significant | | |
| | Abnormal and Clinically significant | | |

# Table. Shift table of Physical examination - Safety population

| | Day 19/ET | | |
|---|---|---|---|
| Screening | Normal | Abnormal and not clinically significant | Abnormal and clinically signficant |
| Normal | | | |
| Abnormal and not clinically significant Abnormal and clinically signficant | | | |

# Table. Vital signs – Safety population

| | | Screening | Baseline | D19/ET | Change from baseline |
|---|---|---|---|---|---|
| Systolic blood pressure (mmHg) | N | | | | |
| | Mean | | | | |
| | SD | | | | |
| | Median | | | | |
| | (Min,Max) | | | | |
| Diastolic blood pressure (mmHg) | | | | | |
| Pulse rate (bpm) | | | | | |
| Vital signs evaluation | N | | | | |
| | Normal | | | | |
| | Abnormal and Not clinically significant | | | | |
| | Abnormal and Clinically significant | | | | |


Table. Shift table of vital signs evaluation – Safety population

| | Day 19/ET | | |
|---|---|---|---|
| Baseline | Normal | Abnormal and not clinically significant | Abnormal and clinically signficant |
| Normal | _ | | |
| Abnormal and not clini significant | ically | | |
| Abnormal and clini signficant | ically | | |

**Table. Ophthalmic examination – Safety population** 

Table. Shift table of ophthalmic examination - Safety population

Table. 12-lead ECG – Safety population

| | | Screening | DAY 19/ET |
|---|---|---|---|
| ECG | N | | |
| | Normal | | |
| | Abnormal and Not clinically significant | | |
| | Abnormal and Clinically significant | | |
| QTC (ms) | N | | |
| | Mean | | |
| | SD | | |
| | Median | | |
| | (Min,Max) | | |
| QTC > 500 ms | N | | |
| | No | | |
| | Yes | | |
| Change in QTC (ms) | N | | |
| | Mean | | |
| Change > 60 ms | N No Yes | | |

Table. Shift table for 12-lead ECG – Safety population




# 9.3.5. Laboratory Parameters

Table. Haematology - Summary statistics - Safety population

| | | Screening | D19/ET | Change from |
|----------------------------|-----------|-----------|--------|-------------|
| | | | | Screening |
| White blood cells (Giga/L) | N | | | |
| | Mean | | | |
| | SD | | | |
| | Median | | | |
| | (Min,Max) | | | |
| ••• | | | | |

 $Table. \ Haematology-Distribution \ by \ normality \ level-Safety \ population$ 

 $Table.\ Haematology-Shift\ table-Safety\ population$ 


Table. Blood chemistry - Summary statistics - Safety population

Table. Blood chemistry – Distribution by normality level – Safety population

Table. Blood chemistry – Shift table – Safety population

Table. Virology at screening – Safety population

Table. Urinalysis \*- Summary statistics - Safety population

\*: only for data in quantitative manner (like pH for exemple)

Table. Urinalysis – Distribution by normality level – Safety population

Table. Urinalysis – Shift table – Safety population

# 9.4. Graphs

Graph. Mean TSS versus time per treatment -PP population

Graph. Median TSS percent change from day 1 by visit and by treatment -PP population

Graph. Mean Erythema versus time per treatment -PP population

Graph. Mean Erythema change from day 1 by visit and by treatment -PP population

Graph. Mean Scaling versus time per treatment -PP population

Graph. Mean Scaling change from day 1 by visit and by treatment -PP population

Graph. Mean Induration versus time per treatment -PP population

Graph. Mean Induration change from day 1 by visit and by treatment -PP population

| 11010 | COI | 110. | ND | ω. | J.DI IX. I |
|--------|-----|------|-------|-----|------------|
| a | | | | | |
| Statis | иcа | ΙÆΙ | iaiy: | 515 | I Iaii |


Graph. Success by visit -PP population

| CCI |
|---------------------------------------------------------------------------|
| Graph. Mean Irritation versus time per treatment -Safety population |
| Graph. Mean Stinging/burning versus time per treatment -Safety population |
| Graph. Mean Pruritus versus time per treatment -Safety population |
| CCI |

Some other descriptive graphics could be performed upon request.





| Internally Approved 01-Feb-2019<br>Protocol No: RD.03.SPR.112075 |
|------------------------------------------------------------------|
| Statistical Analysis Plan |
| CČÍ |
